CLINICAL TRIAL: NCT00583999
Title: Leptin, Soluble Leptin Receptor and Adiponectin in Non Alcoholic Steatohepatitis
Brief Title: The Role of Leptin Receptors in NASH
Acronym: NASH
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 2000513532
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Nonalcoholic Steatohepatitis; Metabolic Syndrome
Keywords: leptin, leptin receptors, adiponectin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Liver biopsy specimes, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: bariatric surgery
  Interventions: Other: no interventions, only regular blood-draw

INTERVENTIONS:
Other: no interventions, only regular blood-draw — No interventions, only regular blood-draw (liver biopsy obtained per routine during the surgery)

SUMMARY:
NAFLD is a spectrum of liver diseases associated with varying degrees of hepatic steatosis, inflammation, and in some cases, fibrosis. NAFLD is a common observation in all demographics, but the prevalence of NAFLD and nonalcoholic steatohepatitis (NASH) is especially high in the morbidly obese population. Leptin is a cytokine that is encoded by the ob gene and primarily secreted by adipose tissue. The production of serum leptin increases with progressive obesity. Because of this observation, there has been significant interest in potential role of leptin in NAFLD.

Our hypothesis is that we will find increased hepatic leptin and leptin receptor expression as the degree of hepatic injury worsens in NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective bariatric surgery, ages 18-65.

Exclusion Criteria:

* non-obese patients, ages less than 18 and over 65. Pregnant patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To link SLR to grade/stage of NASH | 2.5 years

SECONDARY OUTCOMES:
To link SLR, leptin and adiponectin to features/components of the metabolic syndrome | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Torok, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Result] Medici V, Ali MR, Seo S, Aoki CA, Rossaro L, Kim K, Fuller WD, Vidovszky TJ, Smith W, Jiang JX, Maganti K, Havel PJ, Kamboj A, Ramsamooj R, Torok NJ. Increased soluble leptin receptor levels in morbidly obese patients with insulin resistance and nonalcoholic fatty liver disease. Obesity (Silver Spring). 2010 Dec;18(12):2268-73. doi: 10.1038/oby.2010.95. Epub 2010 May 6. PMID 20448542